CLINICAL TRIAL: NCT06692972
Title: Exploration of and Model Establishment of the Regression Pattern of Primary Lesions in Lung Cancer After Definitive Radiotherapy
Brief Title: The Regression Pattern of Primary Lesions in Lung Cancer After Definitive Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Guangying Zhu, Clinical Professor, Chief Physician, China-Japan Friendship Hospital
Other Study IDs: 2024-ZF-38
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; radiotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Definitive radiotherapy is one of the important methods for inoperable locally advanced lung cancer. The recommended dose for definitive radiotherapy is 60-70Gy, and the optimal dose is still uncertain. Residual lesion after radiotherapy is a risk factor for recurrence. High doses to targeted tumor areas can effectively improve the local control rate, while minimizing toxic side effects. The regression pattern of primary lesions in lung caner after radiotherapy has not been clarified. This study intends to retrospectively collect clinical data of lung cancer patients with definitive radiotherapy, and explore the pattern of tumor regression after radiotherapy. It will help optimize the radiotherapy plan for lung cancer, so as to improve the efficacy and prognosis.

DETAILED DESCRIPTION:
This study intends to retrospectively screen and include participants according to inclusion and exclusion criteria, and collect the clinical data of participants by previous medical records. Imaging tools will be used to quantify changes in the spatial location, diameter and volume of target lesions to evaluate tumor regression rate and radiotherapy efficacy, and to explore tumor regression pattern and establish model. In addition, the relationship between tumor regression rate, incidence of adverse radiation events, prognosis and related factors will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Stage II-III lung cancer with a clear pathological diagnosis report or medical record, not undergoing surgery before radiotherapy;
3. The primary lung lesion received definitive radiotherapy (defined as conventional fractionation radiotherapy with dose ≥50Gy, stereotactic radiotherapy with biologically effective dose ≥100Gy);
4. The target lesion of the lung receiving radiotherapy can be measured;
5. Imaging data can be obtained before and after radiotherapy;
6. Complete radiotherapy as planned, or the actual received dose has reached the defined definitive dose.

Exclusion Criteria：

1. Before radiotherapy, the primary lesion of the lung had received local treatment such as surgery or ablative treatment;
2. The radiotherapy plan was not completed, and the actual dose received did not reach the definitive dose (defined as conventional fractionation radiotherapy with dose <50Gy, stereotactic radiotherapy with biologically effective dose <100Gy)；
3. Required imaging data cannot be obtained;
4. Other conditions considered by the investigator to be inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II-III lung cancer patients who have received definitive radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor regression rate | Within 1 year after completion of radiotherapy.
  (1- post-treatment tumor volume/baseline tumor volume)×100%

SECONDARY OUTCOMES:
Objective response rate | Within 1 year after completion of radiotherapy.
  It refers to the proportion of patients who experience a complete or partial remission of tumors in response to treatment, as determined by RECIST criterion.
Disease control rate | Within 1 year after completion of radiotherapy.
  It refers to the proportion of patients who experience an objective response (complete or partial remission) or stable disease in response to treatment, as determined by RECIST criterion.
Progression-free survival | From the start of treatment until the time of disease progression or death, assessed up to 120 months.
  It's calculated from the start of treatment until the time of disease progression or the patient's death, whichever comes first.
Overall survival | From the start of treatment until the time of death, assessed up to 120 months.
  It measures the length of time from the start of treatment until the death of the patient from any cause.
Adverse event rate | Within 1 year after completion of radiotherapy.
  It refers to the frequency of treatment related adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Guangying Zhu, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
Research data including study protocol and statistical analysis plan will be shared after the study is completed and the research results are published.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available starting 1 year and ending 4 years following article publication.
Access Criteria: The data will be made available upon request for researchers who provide a methodologically sound proposal. The data will be accessible for non-commercial research purposes only and will be used to explore additional hypotheses related to the study's objectives.